CLINICAL TRIAL: NCT07324694
Title: Impact of Intraoperative Hemodynamic Instability on Postoperative Major Adverse Events in Cardiac Surgery Patients: A Prospective Cohort Study
Brief Title: Impact of Intraoperative Hemodynamic Instability on Outcomes in Cardiac Surgery
Status: Recruiting | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Osman Uzundere, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: GYTRH-KVC-IOHI-01
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Surgery; Intraoperative Hemodynamic Instability; Postoperative Complication; Acute Kidney Injury; Postoperative Delirium (POD)
Keywords: Intraoperative Hypotension; Cardiopulmonary Bypass; Mean Arterial Pressure; Cohort Study
MeSH Terms: conditions — Postoperative Complications; Acute Kidney Injury; Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodynamic Instability Group: Patients who exhibit intraoperative hemodynamic instability, defined as Mean Arterial Pressure (MAP) < 65 mmHg for >5 minutes continuously, or requiring vasopressor/inotropic support to maintain MAP.
- Hemodynamically Stable Group: Patients who maintain intraoperative hemodynamic stability without significant hypotension episodes (MAP > 65 mmHg) or vasopressor requirement beyond baseline anesthesia induction.

SUMMARY:
Intraoperative hemodynamic instability (IOHI) is a common occurrence during cardiac surgery and is associated with organ hypoperfusion. However, the specific impact of IOHI on composite adverse outcomes remains unclear. This prospective cohort study aims to evaluate the association between intraoperative hemodynamic instability (defined as MAP < 65 mmHg or vasopressor requirement) and major postoperative complications (Delirium, Acute Kidney Injury, Stroke, or Mortality) in adult patients undergoing elective cardiac surgery with cardiopulmonary bypass.

DETAILED DESCRIPTION:
Hemodynamic instability during cardiac surgery is a critical factor influencing postoperative recovery. While transient hypotension is common, prolonged instability may lead to end-organ damage due to hypoperfusion. This prospective observational study will be conducted at the University of Health Sciences Gazi Yasargil Training and Research Hospital.

Patients scheduled for elective cardiac surgery (Coronary Artery Bypass Grafting, Valve replacement/repair, or combined procedures) utilizing cardiopulmonary bypass will be enrolled. Intraoperative hemodynamic data, including Mean Arterial Pressure (MAP), heart rate, and vasoactive medication requirements, will be recorded.

Patients will be categorized into two groups based on intraoperative stability:

1. Hemodynamic Instability Group: Patients experiencing MAP < 65 mmHg for more than 5 minutes continuously or requiring significant vasopressor/inotropic support to maintain target pressure.
2. Stable Group: Patients maintaining hemodynamic stability without significant hypotensive episodes.

The primary endpoint is a composite of major adverse events within 30 days, including Postoperative Delirium (assessed via CAM-ICU), Acute Kidney Injury (KDIGO criteria), Stroke, and All-cause Mortality. Secondary endpoints include the duration of mechanical ventilation and length of ICU/hospital stay. The study aims to provide evidence-based thresholds for intraoperative blood pressure management to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older.
* Scheduled for elective cardiac surgery (CABG, Valve replacement/repair, or combined procedures).
* Surgery performed under cardiopulmonary bypass (CPB).
* Preoperative sinus rhythm.
* Signed informed consent form.

Exclusion Criteria:

* Emergency or salvage surgery.
* Off-pump coronary artery bypass grafting.
* Preoperative mechanical circulatory support (IABP, ECMO) requirement.
* Pre-existing chronic renal failure requiring dialysis (HD/PD).
* Pre-existing cognitive impairment, dementia, or history of psychiatric disorders affecting cooperation.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective cardiac surgery with cardiopulmonary bypass at a tertiary care university hospital.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-04-26 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of Composite Adverse Events | Up to 30 days post-operation
  A composite endpoint defined as the occurrence of any of the following within 30 days post-surgery: Postoperative Delirium (assessed by CAM-ICU), Acute Kidney Injury (KDIGO criteria stage 1 or higher), Stroke (new neurological deficit confirmed by imaging), or All-cause Mortality.

SECONDARY OUTCOMES:
Duration of Mechanical Ventilation | Up to 30 days
  Time from ICU admission to successful extubation (in hours).
Length of Hospital Stay | Up to 30 days
  Total duration of hospital stay from surgery to discharge (in days)
Length of Intensive Care Unit (ICU) Stay | Up to 30 days
  Time from admission to the Intensive Care Unit immediately after surgery until discharge to the ward (in days).

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi Yaşargil Training and Research Hospital, Diyarbakır, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shen X, Tao H, Chen W, Sun J, Jin R, Zhang W, Hong L, Zhang C. Perioperative blood pressure variability as a risk factor for postoperative delirium in the patients receiving cardiac surgery. BMC Anesthesiol. 2024 Nov 25;24(1):424. doi: 10.1186/s12871-024-02817-x. PMID 39581994
- [Result] D'Amico F, Fominskiy EV, Turi S, Pruna A, Fresilli S, Triulzi M, Zangrillo A, Landoni G. Intraoperative hypotension and postoperative outcomes: a meta-analysis of randomised trials. Br J Anaesth. 2023 Nov;131(5):823-831. doi: 10.1016/j.bja.2023.08.026. Epub 2023 Sep 20. PMID 37739903
- [Result] Buitenwerf E, Boekel MF, van der Velde MI, Voogd MF, Kerstens MN, Wietasch GJKG, Scheeren TWL. The haemodynamic instability score: Development and internal validation of a new rating method of intra-operative haemodynamic instability. Eur J Anaesthesiol. 2019 Apr;36(4):290-296. doi: 10.1097/EJA.0000000000000941. PMID 30624247